CLINICAL TRIAL: NCT06962735
Title: Effect of Switching From Intermittently Scanned Continuous Glucose Monitoring to Real-time Continuous Glucose Monitoring on Glycemic Outcomes in Adults With Diabetes: A Real-world, Canadian Retrospective Study
Brief Title: Real-world Effect of Switching From Intermittently-scanned to Real-time Continuous Glucose Monitoring (Switch CGM Retro)
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Switch CGM retro
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- real-time continuous glucose monitoring switch group (rtCGM switch group): adults with diabetes that switched from an isCGM to an rtCGM
  Interventions: Device: real-time continuous glucose monitor
- intermittently scanned continuous glucose monitoring group (isCGM group): adults with diabetes that remained on an isCGM

INTERVENTIONS:
Device: real-time continuous glucose monitor — Individuals who switched from using isCGM to rtCGM
  Groups: real-time continuous glucose monitoring switch group (rtCGM switch group)

SUMMARY:
The objective of this retrospective, observational study, is to better understand the real-world glycemic effectiveness of switching to real time continuous glucose monitoring (rtCGM) from intermittently scanned continuous glucose monitoring (isCGM) among adults with type 1 diabetes or type 2 diabetes in Canada.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older as of the index date
* Clinical diagnosis of T1D or T2D ≥ one year
* Using either MDI or CSII therapy
* Initiated a FreeStyle Libre® isCGM device between January 1, 2018 and July 31, 2023 (isCGM cohort)
* Switched from a FreeStyle Libre® 1 or Libre 2® isCGM device to a Dexcom® G5 or G6 CGM device between April 1, 2018 and July 31, 2023 (rtCGM cohort)
* Baseline HbA1c ≥7.0% for primary objective with rtCGM cohort
* Baseline HbA1c ≥8.0% for key secondary objective comparing rtCGM cohort to isCGM cohort
* Known rtCGM/isCGM start date (month and year)
* Exclusive use of isCGM for ≥ 3 months
* ≥ one HbA1c value up to 6 months (± 6 weeks) prior to index date (HbA1c value must be after isCGM initiation and no more than 6 weeks after the index date)
* ≥ one HbA1c value 6-12 months (± 6 weeks) following the index date
* Informed consent for their medical record data to be used for research purposes

Exclusion Criteria:

* Have a prior history of rtCGM within 12 months of the index date
* Are pregnant at the time of isCGM initiation or time of switch to rtCGM
* Used the isCGM or rtCGM for < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults, who were active patients with type 1 diabetes or type 2 diabetes at LMC, who switched from intermittently scanned continuous glucose monitoring to real-time continuous glucose monitoring (rtCGM switch cohort) or initiated and maintained intermittently scanned continuous glucose monitoring use (isCGM cohort).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c at 6-12-month follow-up compared to baseline | from index date to 6- to-12-month follow-up
  To evaluate change in HbA1c at 6-12-month follow-up compared to baseline after switching from an isCGM system to a rtCGM system in adults with type 1 diabetes

SECONDARY OUTCOMES:
Change in HbA1c in the rtCGM switch cohort compared to a matched isCGM cohort | from index date to 6- to-12-month follow-up
  To compare 6-12 month change in HbA1c in the rtCGM switch cohort, who switched from isCGM to rtCGM, compared to a propensity score matched isCGM cohort, who maintained isCGM use, among a subgroup of patients with T1D and HbA1c ≥ 7.5%.
Change in percent time in target glucose range (TIR) at 6-12 months follow-up | from index date to 6- to-12-month follow-up
  To evaluate change in percent TIR at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in percent time below target glucose range (TBR) | from index date to 6- to-12-month follow-up
  To evaluate change in percent TBR at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in percent time above target glucose range (TAR) | from index date to 6- to-12-month follow-up
  To evaluate change in percent TAR at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in mean glucose | from index date to 6- to-12-month follow-up
  To evaluate change in mean glucose at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in standard deviation (SD) of mean glucose | from index date to 6- to-12-month follow-up
  To evaluate change in SD of mean glucose at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in coefficient of variation (CV) of mean glucose | from index date to 6- to-12-month follow-up
  To evaluate change in CV of mean glucose at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in weight | from index date to 6- to-12-month follow-up
  To evaluate change in weight at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Proportion of patients who achieve HbA1c ≤7.0% | evaluated at 6- to-12-month follow-up
  To evaluate the proportion of patients who achieve HbA1c ≤7.0% at 6-12 months follow-up in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% at baseline and propensity score matched isCGM cohort with HbA1c ≥ 7.5% at baseline.
Weekly incidence of self-reported hypoglycemia | evaluated at 6- to-12-month follow-up
  To evaluate weekly incidence of self-reported hypoglycemia at 6-12 months in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Proportion of patients with ≥ 1 self-reported hypoglycemic event | evaluated at 6- to-12-month follow-up
  To evaluate proportion of patients with ≥ 1 self-reported hypoglycemic event at 6-12 months in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Change in total daily dose (TDD) of insulin | from index date to 6- to-12-month follow-up
  To evaluate change in TDD of insulin at 6-12 months follow-up compared to baseline in the rtCGM switch cohort, and between the rtCGM switch cohort with HbA1c ≥ 7.5% and propensity score matched isCGM cohort with HbA1c ≥ 7.5%.
Proportion of patients using a Tandem® insulin pump in the rtCGM switch cohort | from index date to 6- to-12-month follow-up
  To evaluate proportion of patients using a Tandem® insulin pump in the rtCGM switch cohort during the study period from baseline to 6-12 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a real-world study using data retrieved from a national Diabetes Registry. IPD will not be shared.